CLINICAL TRIAL: NCT07118566
Title: Hyperthermia Combined With Immune Checkpoint Inhibitors in the Treatment of Advanced Gastrointestinal Malignancies With Liver Metastases: A Multicenter, Open-label, Dual-cohort Phase II Exploratory Clinical Study
Brief Title: Hyperthermia Combined With Immune Checkpoint Inhibitors in the Treatment of Advanced Gastrointestinal Malignancies With Liver Metastases
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: China Medical University, China (Other)
Responsible Party: Principal Investigator, Xiujuan Qu, Director, China Medical University, China
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLOG-2025GI-HT01
Record Dates: First submitted 2025-07-28; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-05

CONDITIONS: Gastrointestinal Cancer; Immunotherapy; Liver Metastasis
Keywords: gastrointestinal cancer; immunotherapy; liver metastasis; hyperthermia
MeSH Terms: conditions — Gastrointestinal Neoplasms; Hyperthermia | interventions — Diathermy; Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1: gastric cancer (Experimental): Gastric cancer patients must have received at least one prior line of systemic therapy.
  Interventions: Procedure: Hyperthermia; Drug: Immunotherapy
- Cohort 2: colorectal cancer (Experimental): Colorectal cancer patients must have received at least two prior lines of systemic therapy.
  Interventions: Procedure: Hyperthermia; Drug: Immunotherapy

INTERVENTIONS:
Procedure: Hyperthermia — Each session of hyperthermia should be spaced at least 24 hours apart, with at least one session administered prior to ICI (immune checkpoint inhibitor) treatment. Five times q3w.
  Other Names: Microwave hyperthermia
Drug: Immunotherapy — iv，d1，q3w

SUMMARY:
This study aims to explore the synergistic antitumor effects and safety of hyperthermia combined with immune checkpoint inhibitors (ICIs) in patients with advanced gastrointestinal malignancies with liver metastases. Liver metastasis represents a common cause of treatment failure in gastrointestinal cancers, and the response rate to ICIs remains suboptimal in certain patients with liver metastases, potentially attributable to the immunosuppressive hepatic microenvironment. The combination of hyperthermia with ICIs, chemotherapy, or other therapeutic modalities may further enhance treatment efficacy. Hyperthermia could potentially reverse immunosuppression and improve ICI effectiveness through mechanisms including enhanced tumor blood perfusion, promoted antigen presentation, and increased immune cell infiltration. This multicenter, open-label, dual-cohort phase II trial will evaluate patients stratified by tumor type (colorectal cancer versus gastric cancer) to assess the objective response rate (ORR), progression-free survival (PFS), and safety profile of hyperthermia-ICI combination therapy. Concurrently, dynamic monitoring of peripheral immune markers (such as neutrophil-to-lymphocyte ratio and interleukins) and tumor microenvironment alterations will be conducted to identify potential predictive biomarkers, thereby providing preliminary evidence for subsequent phase III investigations. The ultimate objective is to develop more effective combination treatment strategies for patients with advanced gastrointestinal malignancies accompanied by liver metastases.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years, male or female.
* Histologically or cytologically confirmed diagnosis of gastrointestinal malignancy with liver metastases.
* Prior treatment requirements:

Gastric cancer patients must have received at least one prior line of systemic therapy.

Colorectal cancer patients must have received at least two prior lines of systemic therapy.

* Clinically assessed as suitable for hyperthermia combined with immune checkpoint inhibitor therapy.
* At least one measurable lesion meeting RECIST 1.1 criteria.
* Expected survival ≥6 months.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Adequate organ and bone marrow function.
* Willingness to provide sufficient baseline and post-treatment samples, ability to comply with long-term follow-up and evaluation, and signed informed consent.
* No prior history of other malignancies.

Exclusion Criteria:

* Pregnant or lactating women.
* Any comorbidities or underlying medical conditions that, in the investigator's judgment, render the patient unsuitable for study participation.
* Presence of other severe physical or psychiatric disorders, or clinically significant laboratory abnormalities that may increase the risk associated with study participation, interfere with study results interpretation, or otherwise make the patient inappropriate for inclusion as determined by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2029-05 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | From the start of treatment to tumor progression or death from any cause (whichever occurs first, at least 4 weeks, assessed up to 12 months).
  Objective response rate (ORR) refers to the proportion of patients whose tumor volume has shrunk to the pre-specified value and can maintain the minimum duration requirement (at least 4 weeks, assessed up to 12 months) by the RECIST (Version 1.1), which is the sum of the proportions of complete response (CR) and partial response (PR).

SECONDARY OUTCOMES:
Progression Free Survival | Progression-free survival (PFS) refers to the time from the start of treatment to tumor progression or death from any cause (whichever occurs first, at least 4 weeks, assessed up to 12 months).
Disease Control Rate | From the start of treatment to tumor progression or death from any cause (whichever occurs first, at least 4 weeks, assessed up to 12 months).
  Disease control rate (DCR) refers to the proportion of patients whose tumor volume has shrunk to the pre-specified value and can maintain the minimum duration requirement (at least 4 weeks, assessed up to 12 months) by the RECIST (Version 1.1), which is the sum of the proportions of complete response (CR), partial response (PR), and stable disease (SD).
Overall Survival | From study enrollment through 12 months post-treatment completion of the last participant.